CLINICAL TRIAL: NCT06131827
Title: Combined Effects of Neural Mobilization With Task Based Activities on Spasticity and Motor Function of Upper Limb in Patients With Chronic Stroke.
Brief Title: Neural Mobilization With Task Based Activities on Upper Limb in Patients With Chronic Stroke.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &/23/0233
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Chronic Stroke
Keywords: Neural mobilization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural mobilization (Experimental): Neural mobilization technique will be perormed with twenty oscillations per minute being repeated three sets of one minute respecting one minute interval for rest between each set for 4 days weekly for Six week.
  Interventions: Other: Neural mobilization
- Task based activities (Experimental): Task based activities consisted of different type of task which will be performed with the doasage of 45 minutes per session 5 days weekly for 6 weeks.
  Interventions: Other: Task based activities

INTERVENTIONS:
Other: Neural mobilization — Neural mobilization will be performed with twenty oscillations per minute being repeated three sets of one minute respecting one minute interval of rest between each set for 4 days weekly for six week
  Other Names: Task based activities
  Arms: Neural mobilization
Other: Task based activities — Task based activities consisted of different types task which will be performed with the dosage of 45 minute session 5 days weekly for six week.
  Arms: Task based activities

SUMMARY:
Stroke is defined as sudden neurological disruption of blood supply to brain. It is most common disease that causes severe disabilities like hemiparesis which is most common motor impairment that leads to persistent upper limb dysfunction. In this study we use two techniques to improve upper limb motor dysfunction and reduce spasticity. One is task-based activities which is used to improve motor function and focus on active participation rather than normal movement pattern and other is neural mobilization which aims to reduce spasticity which is most common in stroke patients.

DETAILED DESCRIPTION:
This study will be randomized controlled trial. Participants having stroke past 6 month to 1 year and mini mental state examination score >21 will be included in this study. And participants with severe orthopedic deformity, joint pain and visual impairment will be excluded from this study. The sample size will consist of 34 participants selected through non probability convenient sampling technique, which will further be randomized through sealed envelope method and will divide into two groups .Data will be collected using assessment tools, including the Fugl Mayer assessment scale, box and block test and wolf motor function test. 17 Participants will be assigned to the interventional group (A )which will undergo neural mobilization of median nerve with task based activities .Neural mobilization technique will be performed with twenty oscillations per minute being repeated three sets of one minute respecting one minute interval for rest between each set for 4 days weekly for 6 week.

while task based activities will be performed with the dosage of 45 minutes session 5 days weekly for 6 weeks and 17 participants will be assigned to control group (B

)which will undergo only neural mobilization of median nerve and will receive neural mobilization with twenty oscillations per minute being repeated three sets of one minute respecting one minute interval for rest between each set for 4 days weekly for 6 weeks. After applying both interventions motor function improvement and spasticity reduction will be measured by using BBT, wolf motor scale and fugl -Meyer assessment scale and data will be analyzed through sPss Version 25.

ELIGIBILITY:
Inclusion Criteria:

* Male and female stroke patients.
* 6 month to one year post stroke .
* Age 30-55
* Stable patients
* Mini - mental state examination>2
* Modified ashworth Scale equal<+1

Exclusion Criteria:

* Orthopedic deformity
* Patients undergo bottulinuminjection toxin injection
* Visual impairments
* Joint pain (elbow, shoulder, wrist)

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-22 (Estimated)

PRIMARY OUTCOMES:
Box and block test | 6 weeks
  It measures unilateral gross manual dexterity
Wolf motor Function Test | 6 weeks
  The Wolf Motor Function Test (WMFT) quantifies upper extremity (UE) motor ability through timed and functional tasks
Fugl -Meyer assessment scale | 6 weeks
  It measure motor ability of upper extremity

CONTACTS AND LOCATIONS:
Overall Officials: Memona Ayesha, Ms-NMPT, Principal Investigator — Ripha international university
Locations (1):
- Ripha international university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No